CLINICAL TRIAL: NCT04799808
Title: Investigation of the Immune Response Before and After COVID-19 Disease or SARS-CoV-2 Vaccination in Dialysis Patients, Solid Organ Recipients and Medical Staff
Brief Title: Saxon SARS-CoV-2 Infection and Vaccination Study in Dialysis Patients, Solid Organ Recipients and Staff
Acronym: DIA-Vacc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Universitätsklinikum Leipzig (Other); Klinikum St. Georg gGmbH (Other); Charite University, Berlin, Germany (Other); DRK-Blutspendedienst Nord-Ost gemeinnützige GmbH / Dresden (Unknown); DRK-Blutspendedienst Nord-Ost gemeinnützige GmbH / Institut Plauen (Unknown)
Responsible Party: Principal Investigator, Susanne Dollfus, Prof. Dr. med. Christian Hugo, Technische Universität Dresden
Other Study IDs: DIA-Vacc-21
Record Dates: First submitted 2021-03-08; First posted 2021-03-16 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV-2 Infection; Active Immunization; Immune Response; Immunosuppression
Keywords: SARS-CoV-2; Covid-19; dialysis; immunosuppression; solid organ transplantation; kidney transplant recipients; humoral immimmune response; cellular immune response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples, in particular serum and PBMCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BioNTech cohort: The BioNTech cohort is composed of 1000 study participants who will be protected from SARS-CoV-2 infection by comirnaty vaccine from BioNTech. The study participants consist of mildly immunocompromised dialysis patients, severely immunocompromised solid organ transplant recipients, and the staff caring for them in the nephrology dispensaries.
- Moderna cohort: The Moderna cohort is composed of 1000 study participants who will be protected from SARS-CoV-2 infection by Moderna Biotech vaccine. The study participants consist of mildly immunocompromised dialysis patients, severely immunocompromised kidney transplant recipients, and the staff caring for them in the nephrology dispensaries.

SUMMARY:
To investigate short- (3 and 8 weeks) and long-term (6, 9, 12, and 18 months) immune protection or response at the humoral and cellular levels before and after SARS-CoV-2 infection or vaccination in patients with moderately reduced immune status (dialysis patients) and severely reduced immune status (organ transplant recipients, mostly kidney transplant recipients) and immunocompetent subjects (medical staff) in Saxony, Germany.

DETAILED DESCRIPTION:
* Formation of two separate cohorts of approximately 1000 study subjects each from the three categories (dialysis patients, solid organ transplant recipients and medical staff) of participants vaccinated using either Biontech or Moderna vaccine (Biontech cohort and Moderna cohort, approximately 2000 subjects total).
* Study time points: Before administration of the 1st SARS-CoV-2 vaccine dose, before the 2nd vaccine dose, and 8 weeks and 6, 9, 12, and 18 months after administration of the 1st vaccine dose and after suspected or proven SARS-CoV-2 infection.
* At all time points, a questionnaire or eCRF will be completed with questions about the dialysis center and the clinical course of the patients.
* Humoral immune response will be determined in all study participants.
* Formation of a study subgroup of up to 300 subjects in each cohort (Biontech or Moderna cohort) for detailed evaluation of the cellular immune response (max. 600 subjects in total).
* In case of non-sustained immunity > 6 months as well as the occurrence of a 3rd SARS-CoV-2 infection wave in autumn 2021, this will be investigated analogously to the current wave.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients, organ transplant recipients and medical staff
* written consent to participate in the study

Exclusion Criteria:

* Age < 18 years old

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2000-3000 subjects
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Immune response to SARS-CoV-2 infection or vaccination | 3 to 4 weeks after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Immune response to SARS-CoV-2 infection or vaccination | 8 weeks after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Immune response to SARS-CoV-2 infection or vaccination | 4 months after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Immune response to SARS-CoV-2 infection or vaccination | 6 months after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Immune response to SARS-CoV-2 infection or vaccination | 9 months after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Immune response to SARS-CoV-2 infection or vaccination | 12 months after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Immune response to SARS-CoV-2 infection or vaccination | 15 months after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Immune response to SARS-CoV-2 infection or vaccination | 18 months after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Immune response to SARS-CoV-2 infection or vaccination | 21 months after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Immune response to SARS-CoV-2 infection or vaccination | 24 months after vaccination or infection
  Swab-PCR and/or serological and/or SARS-CoV-2 rapid test proven infection
Humoral response to SARS-CoV-2 infection or vaccination | 3 to 4 weeks after vaccination or infection
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Humoral response to SARS-CoV-2 infection or vaccination | 8 weeks after infection or vaccination
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Humoral response to SARS-CoV-2 infection or vaccination | 4 months after infection or vaccination
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Humoral response to SARS-CoV-2 infection or vaccination | 6 months after infection or vaccination
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Humoral response to SARS-CoV-2 infection or vaccination | 9 months after infection or vaccination
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Humoral response to SARS-CoV-2 infection or vaccination | 12 months after infection or vaccination
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Humoral response to SARS-CoV-2 infection or vaccination | 15 months after infection or vaccination
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Humoral response to SARS-CoV-2 infection or vaccination | 18 months after infection or vaccination
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Humoral response to SARS-CoV-2 infection or vaccination | 21 months after infection or vaccination
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Humoral response to SARS-CoV-2 infection or vaccination | 24 months after infection or vaccination
  SARS-CoV-2 IgA, IgM and different IgG antibody levels
Cellular response to SARS-CoV-2 infection or vaccination | 3 to 4 weeks after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).
Cellular response to SARS-CoV-2 infection or vaccination | 8 weeks after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).
Cellular response to SARS-CoV-2 infection or vaccination | 4 months after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).
Cellular response to SARS-CoV-2 infection or vaccination | 6 months after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).
Cellular response to SARS-CoV-2 infection or vaccination | 9 months after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).
Cellular response to SARS-CoV-2 infection or vaccination | 12 months after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).
Cellular response to SARS-CoV-2 infection or vaccination | 15 months after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).
Cellular response to SARS-CoV-2 infection or vaccination | 18 months after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).
Cellular response to SARS-CoV-2 infection or vaccination | 21 months after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).
Cellular response to SARS-CoV-2 infection or vaccination | 24 months after infection or vaccination
  T cell subtype immunity measured by SARS-CoV-2 interferon-γ release assays (IGRA) and flow cytometry (FC).

SECONDARY OUTCOMES:
SARS-CoV-2 incidence and prevalence | 3 to 4 weeks after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 incidence and prevalence | 8 weeks after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 incidence and prevalence | 4 months after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 incidence and prevalence | 6 months after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 incidence and prevalence | 9 months after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 incidence and prevalence | 12 months after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 incidence and prevalence | 15 months after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 incidence and prevalence | 18 months after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 incidence and prevalence | 21 months after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 incidence and prevalence | 24 months after infection or vaccination
  Survey of the incidence and prevalence of asymptomatic SARS-CoV-2 infections over the study period
SARS-CoV-2 infection or immune response to vaccination | 3 to 4 weeks after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
SARS-CoV-2 infection or immune response to vaccination | 8 weeks after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
SARS-CoV-2 infection or immune response to vaccination | 4 months after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
SARS-CoV-2 infection or immune response to vaccination | 6 months after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
SARS-CoV-2 infection or immune response to vaccination | 9 months after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
SARS-CoV-2 infection or immune response to vaccination | 12 months after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
SARS-CoV-2 infection or immune response to vaccination | 15 months after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
SARS-CoV-2 infection or immune response to vaccination | 18 months after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
SARS-CoV-2 infection or immune response to vaccination | 21 months after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
SARS-CoV-2 infection or immune response to vaccination | 24 months after infection or vaccination
  Differentiation of immunity with respect to SARS-CoV-2 infection versus SARS-CoV-2 vaccination
Strength of immune response | 3 to 4 weeks after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Strength of immune response | 8 weeks after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Strength of immune response | 4 months after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Strength of immune response | 6 months after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Strength of immune response | 9 months after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Strength of immune response | 12 months after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Strength of immune response | 15 months after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Strength of immune response | 18 months after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Strength of immune response | 21 months after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Strength of immune response | 24 months after infection or vaccination
  Assessment of the quantity and specificity of the immune response
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 3 to 4 weeks after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 8 weeks after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 4 months after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 6 months after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 9 months after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 12 months after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 15 months after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 18 months after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 21 months after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
Effect of SARS-CoV-2 vaccination on immune response after asymptomatic disease | 24 months after vaccination
  Influence of vaccination on immunity/immune response in patients with asymptomatic SARS-CoV-2 infection
SARS-CoV-2 vaccination side effects | 3 to 4 weeks after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
SARS-CoV-2 vaccination side effects | 8 weeks after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
SARS-CoV-2 vaccination side effects | 4 months after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
SARS-CoV-2 vaccination side effects | 6 months after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
SARS-CoV-2 vaccination side effects | 9 months after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
SARS-CoV-2 vaccination side effects | 12 months after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
SARS-CoV-2 vaccination side effects | 15 months after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
SARS-CoV-2 vaccination side effects | 18 months after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
SARS-CoV-2 vaccination side effects | 21 months after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
SARS-CoV-2 vaccination side effects | 24 months after vaccination
  Assessing side effects of the different vaccinations in the study cohorts
Effectiveness of vaccination on severity and incidence of COVID-19 | 3 to 4 weeks after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Effectiveness of vaccination on severity and incidence of COVID-19 | 8 weeks after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Effectiveness of vaccination on severity and incidence of COVID-19 | 4 months after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Effectiveness of vaccination on severity and incidence of COVID-19 | 6 months after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Effectiveness of vaccination on severity and incidence of COVID-19 | 9 months after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Effectiveness of vaccination on severity and incidence of COVID-19 | 12 months after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Effectiveness of vaccination on severity and incidence of COVID-19 | 15 months after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Effectiveness of vaccination on severity and incidence of COVID-19 | 18 months after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Effectiveness of vaccination on severity and incidence of COVID-19 | 21 months after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Effectiveness of vaccination on severity and incidence of COVID-19 | 24 months after vaccination or infection
  Assess clinical effectiveness of vaccination (incidence and severity of symptomatic COVID-19 disease)
Duration of vaccination effect | 3 to 4 weeks after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Duration of vaccination effect | 8 weeks after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Duration of vaccination effect | 4 months after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Duration of vaccination effect | 6 months after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Duration of vaccination effect | 9 months after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Duration of vaccination effect | 12 after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Duration of vaccination effect | 15 after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Duration of vaccination effect | 18 months after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Duration of vaccination effect | 21 months after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Duration of vaccination effect | 24 months after vaccination
  Assessment of the duration of an achieved vaccination protection (clinical/immunological)
Compare vaccination effect in different vaccinations and risk populations | 3 to 4 weeks after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Compare vaccination effect in different vaccinations and risk populations | 8 weeks after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Compare vaccination effect in different vaccinations and risk populations | 4 months after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Compare vaccination effect in different vaccinations and risk populations | 6 months after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Compare vaccination effect in different vaccinations and risk populations | 9 months after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Compare vaccination effect in different vaccinations and risk populations | 12 months after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Compare vaccination effect in different vaccinations and risk populations | 15 months after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Compare vaccination effect in different vaccinations and risk populations | 18 months after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Compare vaccination effect in different vaccinations and risk populations | 21 months after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Compare vaccination effect in different vaccinations and risk populations | 24 months after vaccination
  Comparison of vaccination effects/protection in a randomized study cohort with BioNTech vaccine and one with Moderna vaccine
Protection of re-boostering if necessary | 3 to 4 weeks after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)
Protection of re-boostering if necessary | 8 weeks after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)
Protection of re-boostering if necessary | 4 months after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)
Protection of re-boostering if necessary | 6 months after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)
Protection of re-boostering if necessary | 9 months after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)
Protection of re-boostering if necessary | 12 months after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)
Protection of re-boostering if necessary | 15 months after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)
Protection of re-boostering if necessary | 18 months after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)
Protection of re-boostering if necessary | 21 months after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)
Protection of re-boostering if necessary | 24 months after re-boostering
  Assessment of vaccination protection and immune response in case of need for renewed, possibly corrected booster/refresher vaccination in fall 2021 (in case of a 3rd wave and/or in patients with absent or non-sustained vaccination protection)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hugo, Prof., Study Director — Univercity Hospital Carl Gustav Carus
Locations (1):
- Univercity Hospital Carl Gustav Carus, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No